CLINICAL TRIAL: NCT07194499
Title: Knowledge and Attitude Among Healthcare Workers Towards Malaria Vaccine, Sudan 2025.
Status: Completed | Type: Observational
Sponsor: Research and Publication office (Other)
Responsible Party: Sponsor
Other Study IDs: 24008
Record Dates: First submitted 2025-02-09; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-01

CONDITIONS: Malaria; Malaria Vaccine
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No interventions — No intervention

SUMMARY:
This study assesses Sudanese healthcare workers' knowledge and attitudes toward the malaria vaccine in 2025, considering demographic and professional factors. It examines awareness of malaria prevalence, WHO recommendations, vaccine type, efficacy, and safety, along with confidence in recommending it and its acceptability. The findings will aid in designing interventions to improve vaccine uptake and reduce malaria burden.

DETAILED DESCRIPTION:
This study aims to assess the knowledge and attitudes of Sudanese healthcare workers (HCWs) toward the malaria vaccine in 2025. It examines how demographic factors and professional roles influence their understanding and perception. The knowledge assessment includes awareness of malaria prevalence, WHO vaccine recommendations, and vaccine type, efficacy, and safety. The attitude evaluation focuses on confidence in recommending the vaccine and perceptions of its feasibility and acceptance in Sudan. The findings will help design targeted interventions to enhance vaccine uptake and reduce the malaria burden.

ELIGIBILITY:
Inclusion criteria:

* Graduates of healthcare profession fields with at least one year of healthcare practice following graduation.
* Voluntary agreement and written informed consent. exclusion criteria: non medical graduates

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study Population Description:
  The study will include healthcare workers (doctors, nurses, pharmacists, and public health staff) from various healthcare facilities in Sudan.
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2025-01-16 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
Knowledge regarding malaria vaccine | Jan - Apr 2025
  Included 11 questions about awareness, malaria and malaria vaccination
Attitude regarding malaria vaccine | Jan - Apr 2025
  5 point likert-scale assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Research and Publication Office, Khartoum, Khartoum State, Sudan

IPD SHARING:
Plan to Share IPD: No